CLINICAL TRIAL: NCT01008566
Title: A Phase I Trial of Escalating Doses of the Anti-IGF-1R Monoclonal Antibody IMC-A12 and Standard Dose Sorafenib for Treatment of Advanced Hepatocellular Carcinoma
Brief Title: Cixutumumab and Sorafenib Tosylate in Treating Patients With Advanced Liver Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03186; NCI-2012-03186 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHI-64; CCC-PHI-64; 8155; PHI-64 (Other: University of California Davis Comprehensive Cancer Center); 8155 (Other: CTEP); N01CM00038 (NIH); N01CM00071 (NIH); P30CA093373 (NIH)
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Adult Hepatocellular Carcinoma; Advanced Adult Hepatocellular Carcinoma; Localized Non-Resectable Adult Liver Carcinoma; Recurrent Adult Liver Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — cixutumumab; Sorafenib

ARMS (1):
- Treatment (cixutumumab, sorafenib tosylate) (Experimental): Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22 and oral sorafenib tosylate twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cixutumumab; Other: Laboratory Biomarker Analysis; Drug: Sorafenib Tosylate

INTERVENTIONS:
Biological: Cixutumumab — Given IV
  Other Names: Anti-IGF-1R Recombinant Monoclonal Antibody IMC-A12; IMC-A12
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Sorafenib Tosylate — Given orally
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib

SUMMARY:
This phase I trial is studying the side effects and best dose of cixutumumab when given together with sorafenib tosylate in treating patients with advanced liver cancer. Monoclonal antibodies, such as cixutumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving cixutumumab together with sorafenib tosylate may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose (MTD) of IMC-A12 given in conjunction with standard doses of sorafenib to patients with advanced hepatocellular carcinoma (HCC).

II. To describe the toxicity and tolerance of IMC-A12 at each dose studied in combination with standard-dose sorafenib in patients with advanced HCC.

III. To evaluate the impact of IMC-A12 on biomarkers related to the IGF-1R/IGF pathway which is thought relevant to HCC progression and drug resistance.

IV. To obtain preliminary assessments of efficacy through description of progression-free survival (PFS) and objective response rate (RR).

OUTLINE: This is a multicenter, dose-escalation study of cixutumumab followed by an extended accrual phase in which patients are treated at the maximum-tolerated dose.

Patients receive cixutumumab IV over 1 hour on days 1, 8, 15, and 22 and oral sorafenib tosylate twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable or metastatic HCC for which standard curative measures do not exist; the diagnosis of hepatocellular carcinoma should be based on at least one of the following:

  * The presence of one or more liver lesions, measuring ≥ 2 cm, with characteristic arterial enhancement and venous washout in the setting of liver cirrhosis and/or hepatitis B or C infection
  * The presence of liver lesion(s) with AFP >= 400
  * Tissue confirmation in the absence of a and/or b
  * Tissue availability is desired and will be sought, but tissue availability is not mandated for accrual to the study
* No prior systemic therapy for HCC; patients may have had prior embolization, chemoembolization, intra-arterial chemotherapy infusion, ethanol injection, radiofrequency ablation or cryosurgery
* ECOG 0 or 1
* Life expectancy of greater than 3 months
* Absolute neutrophil count > 1,000/mm^3
* Platelets > 65,000/mm^3
* Total bilirubin =< 2 x the institutional upper normal limit
* AST and ALT =< 5 x the institutional upper normal limit
* Renal function =< 1.5 mg/dl or calculated creatinine clearance > 50 mL/min (Cockcroft-Gault formula)
* PT < 4 seconds of prolongation above the upper normal limit
* No evidence of encephalopathy in the last 6 months
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Local therapy for HCC within 4 weeks prior to treatment on this study or those who have not recovered from adverse events related to therapy administered more than 4 weeks earlier
* Receiving other investigational agents
* Brain metastases, because of their poor prognosis, proclivity for progressive neurologic dysfunction that would confound the evaluation of neurologic adverse events, and the potential for increased risk for CNS adverse events
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated on this clinical trial
* HIV-positive patients are ineligible
* Fasting blood glucose > 160 mg/dL
* Esophageal or gastric variceal bleeding within the last 6
* Clinically evident ascites (minimal, medically controlled ascites detectable on imaging studies only is allowed)
* Child-Pugh C cirrhosis or Child-Pugh B cirrhosis with more than 7 points
* Patients unable to swallow the sorafenib tablets whole are ineligible; (the tablets cannot be crushed or broken)
* Cardiac: symptomatic congestive heart failure, unstable angina, clinically significant and uncontrolled cardiac dysrhythmia, uncontrolled hypertension (systolic BP > 150 or diastolic BP > 100 on two occasions within two weeks of beginning therapy on this protocol, myocardial infarction within 6 months, NYHA class > II, LVEF < normal as assessed on MUGA
* Fibrolamellar carcinoma or any mixed variants of HCC with fibrolamellar histology
* Hypersensitivity to human IgG unless the patient has subsequently tolerated IgG agents
* Patients with active hepatitis B infection should be on adequate antiviral therapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-08; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
MTD defined as the highest IMC-A12 dose tested in which none or only one patient had a dose-limiting toxicity (DLT) attributed to IMC-A12 as assessed by NCI CTCAE version 4.0 | First 1 month of therapy
  The toxicities observed at each dose level will be summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity (by CTCAE and nadir or maximum values for the laboratory measures), time of onset (i.e. course number), duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by dose and by course.
Toxicities and tolerability of this regimen as assessed by NCI CTCAE version 4.0 | 30 days

SECONDARY OUTCOMES:
Impact of cixutumumab on biomarkers related to the IGF-1R/IGF pathway | From baseline to up to 5 years
Objective response rate according to RECIST | Up to 5 years
Progression-free rate according to the Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert O'Donnell, Principal Investigator — University of California, Davis
Locations (6):
- United States (6):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Penn State Hershey Cancer Institute-Clinical Trials Office, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania